CLINICAL TRIAL: NCT05456295
Title: Comparative Effect of Carbon Fiber Orthosis Cuff Design on Preference, Comfort, and Mechanics
Acronym: AFOCUFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Fabtech Systems (Unknown)
Responsible Party: Principal Investigator, Jason Wilken, Associate Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 202202450; CDMRP-OP210037 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-06-20; First posted 2022-07-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Lower Limb Injury; Post-Traumatic Osteoarthritis
Keywords: Gait Analysis; Ankle Foot Orthosis; Carbon Fiber; Biomechanics; Adult; Arthritis; Healthy
MeSH Terms: conditions — Leg Injuries; Arthritis

STUDY DESIGN:
Intervention Model Description: All participants will be cast and fit with CDOs with four different proximal cuff designs. CDOs will be labeled as CUFF-A, CUFF-B, CUFF-C, CUFF-D. Testing order of the proximal cuff designs will be randomized to prevent influence of study results.
Who Masked: Participant
Masking Description: Participants will be blinded, to the greatest extent possible, to the different CDO designs and will only be introduced to each device as CUFF-A, CUFF-B, CUFF-C, CUFF-D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- NoCDO (No Intervention): Participants will be tested with no CDO
- CUFF-A (Experimental): The first study CDO will be designated CUFF-A
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- CUFF-B (Experimental): The first study CDO will be designated CUFF-B
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- CUFF-C (Experimental): The first study CDO will be designated CUFF-C
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- CUFF-D (Experimental): The first study CDO will be designated CUFF-D
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)

INTERVENTIONS:
Device: Carbon Fiber Custom Dynamic Orthosis (CDO) — The carbon fiber custom dynamic orthosis will consist of a semi-rigid foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg below the knee. The design of the proximal cuff will differ between CUFF-A, CUFF-B, CUFF-C, CUFF-D.
  Other Names: Ankle Foot Orthosis (AFO)
  Arms: CUFF-A; CUFF-B; CUFF-C; CUFF-D

SUMMARY:
Carbon fiber custom dynamic orthoses (CDOs) consist of a proximal cuff that wraps around the leg just below the knee, a posterior carbon fiber strut that stores and returns energy during gait, and a carbon fiber foot plate that supports the foot and allows bending of the posterior strut. The proximal cuff is a primary interface between the patient and the CDO and may influence comfort, preference, limb mechanics and loading, and effective stiffness of the CDO. The important role of the proximal cuff has not been examined. The purpose of this study is to determine the effects of CDO proximal cuff design on patient reported outcomes, limb mechanics and loading, and CDO mechanical characteristics.

DETAILED DESCRIPTION:
Traumatic lower limb injuries often result in poor functional outcomes with long-term negative effects. Carbon fiber custom dynamic orthoses (CDOs) can improve outcomes by reducing pain, supporting the limb, and transferring forces around the limb through the CDO. CDOs consist of a proximal cuff that wraps around the leg just below the knee, a posterior carbon fiber strut that stores and returns energy during gait, and a carbon fiber foot plate that supports the foot and allows bending of the posterior strut. The proximal cuff is a primary interface between the patient and the CDO and may influence comfort, preference, limb mechanics and loading, and effective stiffness of the CDO. Although CDOs are becoming more commonly prescribed following injury the evidence available to guide clinical practice remains limited. The important role of the proximal cuff has not been systematically examined.

The purpose of this study is to determine the effects of CDO proximal cuff design on patient reported outcomes, limb mechanics and loading, and CDO mechanical characteristics. Two groups of individuals will participate: individuals with post-traumatic osteoarthritis in the ankle and healthy individuals. Testing will occur without an orthosis and while wearing orthoses with four proximal cuff designs representative of currently available devices: 1) a rigid patellar tendon bearing (PTB) clamshell cuff secured using a mechanical ratcheting system, 2) a PTB shell with a fixed pivot point secured with Velcro, 3) a rigid clamshell cuff secured with Velcro, and 4) a semi-rigid cuff with a flexible outer layer secured with Velcro.

ELIGIBILITY:
PARTICIPANTS WITH PTOA:

Inclusion Criteria:

1. Ages 18-65.
2. Diagnosis of ankle PTOA.
3. Ability to walk 50 feet at a slow to moderate pace.
4. Ability to walk without a cane or crutch.
5. Ability to read and write in English and provide written informed consent.

Exclusion Criteria:

1. Diagnosis with a moderate or severe brain injury.
2. Diagnosis with a physical or psychological condition that would preclude functional testing (e.g. cardiac condition, clotting disorder, pulmonary condition…).
3. Ankle weakness as a result of spinal cord injury or nervous system pathology.
4. Nerve, muscle, bone, or other condition limiting function in the contralateral extremity.
5. Rheumatoid or inflammatory arthritis.
6. Necrosis of any bones in the foot or ankle.
7. Pain of 8/10 or greater during walking.
8. Surgery on study limb anticipated in the next 6 months.
9. Uncorrected visual or hearing impairments.
10. Require use of a stabilizing device (i.e. Ankle Foot Orthosis or Knee Orthosis…) to perform daily activities.
11. Pregnancy
12. Body mass index greater than 40.

HEALTHY ABLE-BODIED PARTICIPANTS:

Inclusion Criteria:

1. Ages 18-65.
2. Without current complaint of lower extremity pain, spine pain, open wounds or active infection.
3. Ability to hop without pain.
4. Ability to perform a full squat without pain.
5. Ability to read and write in English and provide written informed consent.

Exclusion Criteria:

1. Diagnosis with a moderate or severe brain injury.
2. Diagnosis with a physical or psychological condition that would preclude functional testing (e.g. cardiac condition, clotting disorder, pulmonary condition).
3. Medical conditions or injuries that have limited participation in work or exercise in the last 6 months.
4. Medical conditions of injuries limiting function for greater than 6 weeks.
5. Uncorrected visual or hearing impairments.
6. Use of an assistive device.
7. Pregnancy
8. Body mass index greater than 35.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Peak Plantar Force (total foot) | Baseline
  Force data (N) collected from the total foot (100% of sensor), measured between the foot and orthosis during gait.
Plantar Force Impulse (total foot) | Baseline
  Plantar force impulse (Ns) across the total foot (100% of sensor) will be calculated using the integral of the force over the stance phase as participants walk in each study condition.
Peak Plantar Force (forefoot) | Baseline
  Force data (N) collected from the total foot (distal 40% of sensor), measured between the foot and orthosis during gait.
Plantar Force Impulse (forefoot) | Baseline
  Plantar force impulse (Ns) across the total foot (distal 40% of sensor) will be calculated using the integral of the force over the stance phase as participants walk in each study condition.
Peak Plantar Force (midfoot) | Baseline
  Force data (N) collected from the total foot (middle 30% of sensor), measured between the foot and orthosis during gait.
Plantar Force Impulse (midfoot) | Baseline
  Plantar force impulse (Ns) across the total foot (middle 30% of sensor) will be calculated using the integral of the force over the stance phase as participants walk in each study condition.
Peak Plantar Force (hindfoot) | Baseline
  Force data (N) collected from the total foot (proximal 30% of sensor), measured between the foot and orthosis during gait.
Plantar Force Impulse (hindfoot) | Baseline
  Plantar force impulse (Ns) across the total foot (proximal 30% of sensor) will be calculated using the integral of the force over the stance phase as participants walk in each study condition.
Numerical Pain Rating Scale | Baseline
  Pain will be assessed using a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable.
PROMIS Patient Reported Outcomes for Physical Function | Baseline
  The Patient Reported Outcome Information System (PROMIS) physical function Computer Adaptive Test (CAT) is a computerized assessment measuring physical function. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents more of the measured variable than the population average.
PROMIS Patient Reported Outcomes for Pain Interference | Baseline
  The Patient Reported Outcome Information System (PROMIS) pain interference Computer Adaptive Test (CAT) is a computerized assessment measuring pain interference. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents more of the measured variable than the population average.
Participant Device Preference | Baseline
  The participant will rank order their preference for their standard of care device (if applicable), NoCDO, CUFF-A, CUFF-B, CUFF-C, CUFF-D on a questionnaire.

SECONDARY OUTCOMES:
Ankle Range of Motion | Baseline
  Peak ankle dorsiflexion (degrees) during gait.
Peak Ankle Moment | Baseline
  Peak ankle moment (Nm/kg) during gait.
Peak Ankle Power | Baseline
  Peak ankle power (W/kg) during gait.
Modified Socket Comfort Score (Comfort) | Baseline
  Comfort scores range from 0 = most uncomfortable to 10 = most comfortable.
Modified Socket Comfort Score (Smoothness) | Baseline
  Comfort scores range from 0 = least smooth to 10 = most smooth.

OTHER OUTCOMES:
Center of Pressure Velocity Timing | Baseline
  Timing of peak center of pressure velocity (percent stance) during gait.
Center of Pressure Velocity Magnitude | Baseline
  Magnitude of peak center of pressure velocity (m/s) during gait.
Tibialis Anterior Muscle Activity | Baseline
  Electromyography (EMG, % Maximum) of the tibialis anterior during gait.
Peroneus Longus Muscle Activity | Baseline
  Electromyography (EMG, % Maximum) of the peroneus longus during gait.
Soleus Muscle Activity | Baseline
  Electromyography (EMG, % Maximum) of the soleus during gait.
Medial Gastrocnemius Muscle Activity | Baseline
  Electromyography (EMG, % Maximum) of the medial gastrocnemius during gait.
Semi-Structured Interview | Baseline
  Semi-structured interviews will also be used to fully capture the patients' perspectives, experience, and opinions associated with the device options they experienced as part of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilken, PT, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No